CLINICAL TRIAL: NCT03061175
Title: Facilitating Informed Decisions for Contralateral Prophylactic Mastectomy
Brief Title: Web-Based Decision Aid in Improving Informed Decisions in Patients With Stage 0-IIIA Breast Cancer Considering Contralateral Prophylactic Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sharon Manne, PhD, Professor of Medicine, Rutgers Cancer Institute of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro20150001914; NCI-2017-00173 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro20150001914; 131504 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH); R21CA187643 (NIH)
Record Dates: First submitted 2017-02-13; First posted 2017-02-23 (Actual); Results first posted 2020-07-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Stage 0 Breast Cancer; Stage I Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer
MeSH Terms: conditions — Breast Carcinoma In Situ; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Web-Based Contralateral Prophylactic Mastectomy CPM-DA) (Experimental): Patients receive a website address, a secure username and password, and instructions for using the web-based Contralateral Prophylactic Mastectomy (CPM)- Decision Aid (DA).
  Interventions: Other: Internet-Based Intervention; Other: Survey Administration
- Arm II (Usual Care) (Experimental): Patients undergo usual care available to patients considering CPM and receive information from a medical oncologist about CPM.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Internet-Based Intervention — Receive web-based CPM-DA
  Arms: Arm I (Web-Based Contralateral Prophylactic Mastectomy CPM-DA)
Other: Survey Administration — Ancillary studies

SUMMARY:
This pilot randomized clinical trial studies how well a web-based decision aid works in improving informed decisions in patients with stage 0-IIIA breast cancer considering contralateral prophylactic mastectomy (CPM). A web-based decision aid (DA) may help doctors determine how patients make decisions about whether or not to have contralateral prophylactic mastectomy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop a feasible web-based decision aid (DA).

SECONDARY OBJECTIVES:

I. To provide preliminary data on the impact of the contralateral prophylactic mastectomy (CPM)-DA on preparedness to make the CPM decision, decisional conflict, CPM knowledge, psychosocial factors, perceived risk for cancer in the healthy/breast/metastatic disease, cancer recurrence/metastasis worry, cancer distress and intention to have CPM.

OUTLINE:

PHASE I (PROTOTYPE DEVELOPMENT AND TESTING): Patients attend an interview and are asked questions about experiences with CPM, reasons they chose and did not choose CPM, and CPM satisfaction for 60 minutes. Patients then receive access to web-based CPM-DA and attend an interview over 90 minutes to provide feedback on module and to complete a prototype evaluation.

PHASE II (CPM-DA FEASIBILITY TRIAL): Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo usual care (UC) available to patients considering CPM and receive information from a medical oncologist about CPM.

ARM II: Patients receive a website address, a secure username and password, and instructions for using the web-based CPM-DA.

After completion of study treatment, patients are followed up at 2-4 weeks and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* PHASE I: Has a first, primary diagnosis of unilateral stage 0, 1, 2, or 3a breast cancer (patients with bilateral breast cancer will be excluded from participation)
* PHASE I: Speaks and reads English
* PHASE I: Women with sporadic cancers (WSC) (does not have hereditary breast/ovarian cancer syndrome [BReast CAncer gene (BRCA) carrier, strong family history]); if there is any uncertainty, the surgeon will use the Tyrer-Cuzick (Tyrer et al., 2004) risk model to calculate risk; the Tyrer-Cuzick model calculates a personal lifetime risk of breast cancer based on multiple factors; it has become the standard model because it incorporates not only factors such as estrogen exposure and first degree relatives, but also second degree relatives and paternal lineage; a lifetime risk of 20% or greater is considered high risk and would necessitate increased screening methods to the traditional annual mammogram; for this study, anyone with a lifetime risk up to 19% on the Tyrer-Cuzick model will be considered average risk for breast cancer; anyone with a lifetime risk of 20% or greater will be excluded from participation
* PHASE I: Able to provide meaningful informed consent
* PHASE II: Completed initial surgical consult with breast cancer surgeon at Cancer Institute of New Jersey (CINJ)/Massachusetts General Hospital (MGH)/Memorial Sloan Kettering Cancer Center (MSKCC) and is considering CPM, regardless of the surgical treatment of their primary breast cancer (lumpectomy/mastectomy)
* PHASE II: Has home internet access
* PHASE II: Has a first, primary diagnosis of unilateral stage 0, 1, 2, or 3a breast cancer
* PHASE II: Speaks and reads English
* PHASE II: WSC (does not have hereditary breast/ovarian cancer syndrome [BRCA carrier, strong family history]); if there is any uncertainty, the surgeon will use the Tyrer-Cuzick (Tyrer et al., 2004) risk model to calculate risk; for this study, anyone with a lifetime risk up to 19% on the Tyrer-Cuzick model will be considered average risk for breast cancer; anyone with a lifetime risk of 20% or greater will be excluded from participation
* PHASE II: Able to provide meaningful informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-09-24 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Manne, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Web-Based Contralateral Prophylactic Mastectomy CPM-DA): Patients receive a website address, a secure username and password, and instructions for using the web-based Contralateral Prophylactic Mastectomy (CPM)-Decision Aid (DA).
  Internet-Based Intervention: Receive web-based CPM-DA
  Survey Administration: Ancillary studies
- Arm II (Usual Care): Patients undergo usual care available to patients considering Contralateral Prophylactic Mastectomy (CPM) and receive information from a medical oncologist about CPM.
  Survey Administration: Ancillary studies
Period: Baseline
Arm/Group | Arm I (Web-Based Contralateral Prophylactic Mastectomy CPM-DA) | Arm II (Usual Care)
Started | 47 | 47
Completed | 46 | 47
Not Completed | 1 | 0
Not completed — Participant was deemed ineligible | 1 | 0
Period: Followup 1 at 2-4 Weeks Post-surgery
Arm/Group | Arm I (Web-Based Contralateral Prophylactic Mastectomy CPM-DA) | Arm II (Usual Care)
Started | 45 (1 Participant dropped out of the study before the follow-up survey was to be sent) | 47
Completed | 39 (39 participants completed the follow-up survey out of the 45 who were sent the survey) | 44 (44 participants completed the follow-up survey out of the 47 who were sent the survey)
Not Completed | 6 | 3
Not completed — Skipped assessment | 6 | 2
Not completed — Withdrawal by Subject | 0 | 1
Period: Followup 2 at 6 Months
Arm/Group | Arm I (Web-Based Contralateral Prophylactic Mastectomy CPM-DA) | Arm II (Usual Care)
Started | 45 (Participants who skipped the first follow-up survey were still sent the second FU survey) | 46 (1 participant withdrew from the study in between the 1st and 2nd follow-up survey so only 46 sent)
Completed | 41 (41 participants completed the 2nd follow-up survey out of the 45 who were sent the survey) | 39 (39 participants completed the follow-up survey out of the 46 who were sent the survey)
Not Completed | 4 | 7
Not completed — Lost to Follow-up | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Arm I (Web-Based CPM-DA): Patients receive a website address, a secure username and password, and instructions for using the web-based CPM-DA.
  Internet-Based Intervention: Receive web-based CPM-DA
  Survey Administration: Ancillary studies
- Total: Total of all reporting groups
Arm/Group | Arm I (Web-Based CPM-DA) | Arm II (Usual Care) | Total
Number analyzed (Participants) | 46 | 47 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] — Age reported as Mean with Standard Deviation
  years | 47.5 (8.4) | 45.5 (8.4) | 46.5 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants] — All participants are female per inclusion criteria.
  Participants
    Female | 46 | 47 | 93
    Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was collected as Hispanic/Latino (Yes or No) Race was collected as Caucasian, African American, Asian, Hawaiian/Pacific Islander, American Indian/Alaskan Native, Two or more races, unknown/not reported
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 2 | 3 | 5
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 4 | 6
    White | 39 | 35 | 74
    More than one race | 2 | 1 | 3
    Unknown or Not Reported | 0 | 4 | 4
Education [Count of Participants; unit: Participants] — Education was categorized as high school, Some college, Tech or Trade School, college graduate, some graduate work, and graduate degree.
  Participants
    High school | 2 | 3 | 5
    Some college | 8 | 6 | 14
    Tech or trade school | 1 | 1 | 2
    College Graduate | 15 | 17 | 32
    Some Graduate Work | 2 | 3 | 5
    Graduate Degree | 18 | 17 | 35
Recruitment Site [Count of Participants; unit: Participants] — Site participant was recruited from
  Participants
    MSKCC | 36 | 37 | 73
    MGH | 10 | 10 | 20
Marital Status [Count of Participants; unit: Participants] — Marital status was characterized as Married, Single, Divorced/Widowed
  Participants
    Married | 38 | 36 | 74
    Single | 5 | 7 | 12
    Divorced/Widowed | 3 | 4 | 7
Employment Status [Count of Participants; unit: Participants] — Employment Status was categorized as Full Time, Part Time, On leave, Does not work
  Participants
    Full Time | 28 | 23 | 51
    Part Time | 8 | 9 | 17
    On Leave | 5 | 4 | 9
    Does not work | 5 | 11 | 16
Income [Count of Participants; unit: Participants] — Income was categorized as <$60,000, $60-$139,999, $140,000-$179,999,
  >$180,000 or missing
  Participants
    < $60,000 | 7 | 10 | 17
    $60,000-$139,999 | 17 | 17 | 34
    $140,000-$179,999 | 5 | 6 | 11
    >$180,000 | 14 | 10 | 24
    missing | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Contralateral Prophylactic Mastectomy (CPM) Knowledge Assessed by Surveys for CPM-DA Participants vs. UC Participants
Description: CPM knowledge is a 10-item multiple-choice measure developed by author Kirsten and Smith. Scores range from 0-100% correct with a higher score equaling more correct knowledge items. Items assessed understanding of the definition of CPM, surgical recovery time and risks/side effects, whether or not CPM improves survival, and whether CPM reduced the risk for disease progression. Will characterize the data using standard methods (estimated marginal means, standard errors, and Cohen's d effect sizes) separately by study arm. At follow-up scores will be reported as the difference between the knowledge score at two time points- the baseline knowledge score and follow-up knowledge score for both the CPM-DA arm and the UC arm.
Time Frame: 2-4 week follow up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm I (Web-Based CPM-DA) | Arm II (Usual Care)
Number analyzed (Participants) | 39 | 44
score on a scale | 62.47 (3.40) | 51.33 (3.24)

2. Primary Outcome: Preparedness to Make the Contralateral Prophylactic Mastectomy Decisions as Assessed by Surveys
Description: Preparedness for the CPM decision was assessed using a 16-item scale adapted from the Ottawa Preparation for Decision Making scale modified to address the CPM decision. Items evaluated the amount of and satisfaction with information about CPM. Scores were reported as a mean across the items and ranged from 1-4 with 1 = Strongly Disagree; 2= Moderately Disagree; 3 = Moderately Agree; 4= Strongly Agree Higher scores = more prepared. Outcomes reported as estimated marginal means, standard errors, and effect size measures for usual care and B-Sure decision aid conditions.
Time Frame: 2-4 week follow up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm I (Web-Based CPM-DA) | Arm II (Usual Care)
Number analyzed (Participants) | 39 | 44
score on a scale | 3.46 (.09) | 3.42 (.08)

3. Primary Outcome: Decisional Conflict Assessed by the Decisional Conflict Scale
Description: The Ottawa Decisional Conflict scale has 16 items and five subscales: support for the decision, uncertainty about the decision, level of relevant information, clarity of relevant values, and effective decision. Items are rated on a 5-point Likert scale (0= Strongly Disagree to 4 = Strongly Agree). Scores for the five subscales were calculated by an average that was multiplied by 25, which is recommended by the scale's developers. Thus, scores can range from 0 (no decision conflict) to 100 (high decision conflict). Higher scores indicate more decisional conflict.
Time Frame: 2-4 week follow up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm I (Web-Based CPM-DA) | Arm II (Usual Care)
Number analyzed (Participants) | 39 | 44
score on a scale
  Uncertainty | 26.38 (3.50) | 25.51 (3.23)
  Informed | 13.43 (1.96) | 17.13 (1.81)
  Values Clarity | 15.50 (2.05) | 20.76 (1.90)
  Support | 12.48 (2.51) | 16.33 (2.33)
  Effective Decision | 9.65 (1.90) | 12.46 (1.77)
  Confidence in Decision | 9.10 (0.35) | 8.50 (0.33)

4. Secondary Outcome: Self-Efficacy at 2-4 Week Follow up Survey
Description: Self-efficacy was a 3-item measure of confidence in the ability to manage worries and uncertainty about a possible recurrence of breast cancer, concerns about future surveillance, and worries about undergoing future surveillance. Results reported as Estimated marginal means, standard errors, and effect size measures for usual care and B-Sure decision aid conditions. Scores were reported as the mean across the 3 items and ranged from 1 = Not at all confident; 2 = Somewhat confident; 3 = Moderately confident; 4 = Very confident; 5 = Extremely confident. Higher scores indicate more self-efficacy.
Time Frame: 2-4 week follow up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm I (Web-Based CPM-DA) | Arm II (Usual Care)
Number analyzed (Participants) | 39 | 44
score on a scale | 4.00 (0.16) | 3.85 (.014)

5. Secondary Outcome: Cancer Worry Assessed by 2-4 Week Follow-up Surveys
Description: Worry is measured by a single item that asks how worried the participant is about having another form of breast cancer on a four-point Likert scale 1= not at all worried and 4 = very worried. Higher scores indicate more worry. Results reported as estimated marginal means, standard errors, and effect size measures for usual care and B-Sure decision aid conditions
Time Frame: 2-4 week follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm I (Web-Based CPM-DA) | Arm II (Usual Care)
Number analyzed (Participants) | 39 | 44
score on a scale | 2.91 (0.24) | 2.84 (0.21)

6. Secondary Outcome: CPM Motivations Assessed by Surveys
Description: Reasons for CPM were measured by an 11-item scale developed after a review of the qualitative and quantitative literature on motivations for CPM and interviews with women who chose or did not choose CPM. Scored were reported as a mean score across the 11 items. The scale was scored on a 1-4 scale from not at all important to Yes, extremely important and Higher score = more reasons/motivations. Outcomes reported as Estimated marginal means, standard errors, and effect size measures for usual care and B-Sure decision aid conditions
Time Frame: 2-4 week follow up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm I (Web-Based CPM-DA) | Arm II (Usual Care)
Number analyzed (Participants) | 39 | 44
score on a scale | 2.77 (0.12) | 2.73 (0.11)

7. Secondary Outcome: Perceived Risk of Recurrence Assessed by 2 Items on Surveys
Description: Perceived risk was measured by two items. One item assessed contralateral breast cancer risk risk after unilateral mastectomy and radiation. The second item assessed perceived risk for chest wall recurrence after CPM. The first item asked "Out of 100 women with early breast cancer are treated with a single mastectomy or lumpectomy and radiation, about how many will develop breast cancer in the "other breast" in the 5 years after treatment? ___ women out of 100". The second item assessed risk for chest wall recurrence after bilateral mastectomy using the same scale 2. "If 100 women with early breast cancer have both breasts removed, how many will have breast cancer come back in the chest wall area of the "other breast" in the five years after treatment?". Outcomes reported as Estimated marginal means and standard errors for usual care and B-Sure decision aid conditions of the # out of 100 that women reported.
Time Frame: 2-4 week follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm I (Web-Based CPM-DA) | Arm II (Usual Care)
Number analyzed (Participants) | 39 | 44
score on a scale
  Risk for CBC after unilateral mastectomy/Radiation | 6.44 (1.97) | 5.10 (1.98)
  risk for chest wall recurrence | 11.95 (2.52) | 12.12 (2.26)

8. Other Pre Specified Outcome: User Interface Satisfaction Survey
Description: The scale has 27 items and four subscales: usefulness, ease of use, ease of learning, and satisfaction. Scales ranged from 1-7 with 1 being not at all or strongly disagree up to 7 being definitely or strongly agree.
Time Frame: 2-4 week follow up
Population: Results provided for B-sure intervention arm only as usual care did not view or evaluate B-sure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Web-Based CPM-DA) | Arm II (Usual Care)
Number analyzed (Participants) | 37 | 0
score on a scale
  Overall Evaluation | 5.63 (0.77) |
  Usefulness | 4.92 (1.42) |
  Ease of use | 6.03 (0.76) |
  Ease of learning | 6.21 (0.96) |
  Satisfaction | 5.56 (1.52) |

9. Other Pre Specified Outcome: B-Sure Use- Time
Description: Basic descriptive information will be gathered regarding the length of time modules are viewed. B-Sure use will be assessed by average time spent in B-Sure
Time Frame: 2-4 week follow up
Population: Data reported is for participants in the B-Sure intervention arm only. The usual care participants did not receive the intervention.
Measure: Mean (Full Range); unit: Minutes
Arm/Group | Arm I (Web-Based CPM-DA) | Arm II (Usual Care)
Number analyzed (Participants) | 37 | 0
Minutes | 52.68 [2 to 107] |

ADVERSE EVENTS:
Time Frame: 6 Months.
Description: For the purposes of this study, an adverse event was defined as a participant experiencing any psychological distress, as reported by the patient to the study staff.
Arm/Group | Arm I (Web-Based CPM-DA) | Arm II (Usual Care)
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/47
Other Adverse Events (participants affected / at risk) | 0/46 | 1/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Web-Based CPM-DA) (N=46) | Arm II (Usual Care) (N=47)
Participant reported distress to study staff (Social circumstances) | 0 (0) | 1 (1) — Participant reported distress to study staff

LIMITATIONS AND CAVEATS:
Future studies would benefit from a larger randomized trial including more minorities, lower education & income, & patients seen in community-based settings

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT03061175/Prot_SAP_001.pdf
  • Informed Consent Form (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT03061175/ICF_000.pdf